CLINICAL TRIAL: NCT03961789
Title: Assessment of the Satisfaction of Patient Undergoing Opioid Replacement Therapy Toward Their Management in Community Pharmacy - SATISFY: a Cross-sectional Study
Brief Title: Assessment of the Satisfaction of Patient Undergoing Opioid Replacement Therapy Toward Their Management in Community Pharmacy
Acronym: SATISFY
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UFR de Pharmacie (Clermont-Ferrand) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-434
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid-Related Disorders; Opiate replacement therapy; Community Pharmacy Services; Patient Satisfaction
MeSH Terms: conditions — Opioid-Related Disorders; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohorte 1: patients undergoing opioid replacement therapy
  Interventions: Other: patients undergoing opioid replacement therapy

INTERVENTIONS:
Other: patients undergoing opioid replacement therapy — patients undergoing opioid replacement therapy
  Other Names: no intervention or other

SUMMARY:
The patient's compliance to his medication therapy, and therefore the success of the treatment, is particularly related to his pharmacy management. Thus, the satisfaction of an individual in their interview with the pharmacist is a very important element.

The pharmacist in his professional activity may have to manage patients with opioid related disorders. Pharmacist activity will result in the dispensing of opioid replacement therapy (ORT), single-use syringes, harm reduction kits and prevention advices for the reduction of toxicity and infection risks.

Since the 1990s, the consumption of ORT has been steadily increasing. According to the OFDT (French Observatory of Drugs and Drug Addiction), the number of patients undergoing ORT is about 150 000 patients. Since high-dose buprenorphine is prescribed for approximately two-thirds of patients, it remains the most frequently prescribed ORT in France.

Recently, a French association assisting drug users (ASUD - Auto-support des usagers de drogues) performed a study in Paris (20/07/2018 - 25/08/2018) to assess the delivery of opioid replacement therapies by community pharmacists. In this study, 71% of pharmacists refused to deliver opioid replacement therapies. The main reasons reported were security (56%) and activity saturation, meaning that pharmacists considered that they had too many patients using opioid drugs. In France, the refusal of a pharmacist to deliver drugs is a punishable offence. According to the Code of ethics of pharmacists, pharmacists must respect life and people without discrimination. Pharmacists have a low perception of patients suffering from opioid addiction. Another study performed by ASUD in 93 community pharmacies, showed that pharmacists used the term "toxicomaniacs" instead of "drug users". Most pharmacists had had a bad experience with drugs users, with physical and verbal aggressions. The conclusions of this study showed that pharmacists lacked knowledge of drug users and drug use. Pharmacists knew about harm reduction kits for opioid users (containing sterile syringes, needles, water, antiseptics, etc.) and had already opened them, but very few knew how to use them. More worryingly, some pharmacists did not understand the harm reduction strategies available It thus appears that community pharmacists have a difficult relationship with patient suffering of opioid related disorders, which can have an impact on patient's satisfaction.

The objective of this study will be to assess the satisfaction of patients undergoing ORT regarding their management by community pharmacists.

DETAILED DESCRIPTION:
Patients will be recruited in addiction departments, associations for risk management and general practitioners, and a paper questionnaire will be sent to the patients. The questionnaire is anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing opioid replacement therapy

Exclusion Criteria:

* Age <18 years
* Patient unable to understand or write in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing opioid replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Score of satisfaction | day 1
  visual analogic scale (VAS) "Are you satisfied with your management by community pharmacists?" 0: not satisfied - 100: totally satisfied

SECONDARY OUTCOMES:
Prevention tips given by the pharmacist: risk of infection, overdose, way of using drugs, adverse effects and drug interactions | day 1
  yes/no
Services rendered by the pharmacist: sale of sterile equipment, management of soiled waste, dispensing of opioid replacement therapy | day 1
  yes/no
Perception of the profile / behaviour of pharmacists: welcoming and open to discussion | day 1
  VAS, 0: not at all - 100 : totally
Perception of the profile / behaviour of pharmacists: respect for confidentiality | day 1
  VAS, 0: not at all - 100 : totally
Perception of the profile / behaviour of pharmacists: competent | day 1
  VAS, 0: not at all - 100 : totally
opioid replacement therapy | day 1
  name, dose, route
Number of physician consulted for the last 6 months | day 1
  number
Number of community pharmacy consulted for the last 6 months | day 1
  number
duration of opioid use disorder | day 1
  number of years/months
Demographic information | day 1
  : age, sex, study level, marital status, health care insurance, monthly income, type of housing

CONTACTS AND LOCATIONS:
Overall Officials: David Balayssac, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France